CLINICAL TRIAL: NCT05219864
Title: Topical Ruxolitinib Evaluation in Chronic Hand Eczema Study 1 (TRuE-CHE1): A Phase 3, Double-Blind, Randomized, 16-Week, Vehicle-Controlled, Efficacy and Safety Study of Ruxolitinib Cream Followed by an Open-Label Extension Period in Adults With Chronic Hand Eczema
Brief Title: Topical Ruxolitinib Evaluation in Chronic Hand Eczema Study 1
Acronym: TRuE-CHE1
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision; no safety concerns.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-313
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Hand Eczema
Keywords: eczema; chronic hand eczema (CHE); dermatitis; skin disease; JAK inhibitor
MeSH Terms: conditions — Eczema; Dermatitis; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Participants will receive ruxolitinib cream (1.5%) or vehicle cream for 16 weeks, after which they will be offered the opportunity to receive ruxilitinib cream (1.5%) in the open-label treatment extension period for another 16 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib (Experimental): Ruxolitinib cream 1.5% twice daily (BID) for 16 weeks followed by ruxolitinib cream 1.5% BID for an additional 16-week treatment extension period.
  Interventions: Drug: Ruxolitinib cream
- Vehicle (Placebo Comparator): Vehicle cream for 16 weeks followed by crossover to ruxolitinib cream 1.5% BID in a 16-week treatment extension period.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB18424 cream
  Arms: Ruxolitinib
Drug: Vehicle — Vehicle cream is a topical formulation applied as a thin film to affected areas.
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib cream in adult participants with diagnosis of chronic hand eczema (CHE) and moderate to severe disease activity (Investigator's Global Assessement (IGA) of CHE score 3 or 4).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chromic hand eczema (CHE) as defined by hand eczema (HE) lasting > 3 months or ≥ 2 flares within the previous 12 months.
* Screening and baseline IGA-CHE 3 or 4.
* Baseline CHE-related Itch NRS ≥ 4.
* Recent history (within the past 1 year of baseline) of inadequate response to treatment with topical corticosteroids (TCS), topical calcineurin inhibitors (TCI), or oral alitretinoin; or intolerance or contraindication to TCS or TCI or oral alitretinoin.
* Willingness to avoid pregnancy or fathering children based on the criteria below.

Exclusion Criteria:

* Known triggers for CHE (allergic or irritant, such as those identified by previous patch tests) cannot be avoided during the course of this study.
* Participants who have an unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to baseline.
* Participants with concurrent conditions and history of other diseases such as other active skin disease or infection on the hands; immunocompromised; chronic or acute infection requiring systemic treatments; active acute skin infection; other concomitant skin conditions that may interfere with study assessments or compromise participant safety; other types of eczema; chronic asthma requiring high dose of inhaled corticosteroids; current or history of hepatitis B or C virus infection.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Laboratory values outside of the protocol-defined criteria.
* Use of protocol-defined treatments within the indicated washout period before baseline.
* Psoralen ultraviolet A (PUVA) or ultraviolet B (UVB) therapy on the hands within 4 weeks before baseline.
* Pregnant or lactating participants, or those considering pregnancy during the period of their study participation.
* Further exclusion criteria apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2024-04-25 (Estimated); Study Completion 2024-09-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving Investigator's Global Assessment-Chronic Hand Eczema Treatment Success (IGA-CHE-TS) | Week 16
  The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). IGA-CHE treatment success (IGA-CHE TS) is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from baseline.

SECONDARY OUTCOMES:
Proportion of participants with a ≥ 4-point improvement in chronic hand eczema (CHE) related Itch NRS score | Week 16
  The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and subject will rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable) on a daily basis.
Proportion of participants with a ≥ 2-point improvement in CHE-related Pain NRS score | Week 16
  The Pain NRS is a validated, self-reported, instrument for measurement of itch intensity and subject will rate the intensity of their pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Change from baseline in the modified Total Lesion Symptom Score (mTLSS) | Up to Week 32
  The mTLSS is a validated tool for assessing hand eczema. The scale quantifies the 7 features (erythema, scaling, hyperkeratosis/lichenification, vesiculation, oedema, fissures, and pruritus/pain) of HE (0 = none, 1 = mild, 2 = moderate, and 3 = severe).
Proportion of participants achieving an IGA-CHE-TS from baseline | Up to Week 32
  The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). IGA-CHE treatment success (IGA-CHE TS) is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from baseline.
Change from baseline in CHE-related Itch Numerical Rating Scale (NRS) score (weekly average) | Up to Week 32
  The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and subject will rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable).
Change from baseline in CHE-related Pain NRS score (weekly average) | Up to Week 32
  The Pain NRS is a validated, self-reported, instrument for measurement of itch intensity and subject will rate the intensity of their pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Time to ≥ 4-point improvement from baseline in CHE-related Itch NRS score | Up to Week 32
  The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and subject will rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable) on a daily basis.
Time to ≥ 2-point improvement from baseline in CHE-related Pain NRS score. | Up to Week 32
  The Pain NRS is a validated, self-reported, instrument for measurement of itch intensity and subject will rate the intensity of their pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable) on a daily basis.
Percentage change in Hand Eczema Severity Index (HECSI) | Week 16
  The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales.
Proportion of Participants with HECSI-75 | Weeks 2, 8, 16 and 32
  HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales.
Proportion of participants with HECSI-90 | Weeks 2, 8, 16, and 32
  HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales.
Mean Patient Global Impression of Change (PGIC) score | Up to Week 32
  The Patient Global Impression of Change (PGIC)is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Proportion of participants with each score on the PGIC | Up to Week 32
  The PGIC is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Proportion of Participants with a score of either 1 or 2 on the PGIC | Up to Week 32
  The PGIC is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Haq Nawaz, MD, Study Director — Incyte Corporation
Locations (49):
- United States (26):
  - Southwest Skin Specialists Phoenix Biltmore, Phoenix, Arizona
  - Raoof Md Encino, Encino, California
  - First Oc Dermatology, Fountain Valley, California
  - Marvel Clinical Research Llc, Huntington Beach, California
  - Well Pharma Medical Research Corporation, Miami, Florida
  - Psoriasis Treatment Center of South Florida, Pembroke Pines, Florida
  - Lenus Research Medical Group, Llc, Sweetwater, Florida
  - Delricht Research, Marietta, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Midwest Allergy Sinus Asthma, Sc, Springfield, Illinois
  - Dermatologist Specialist, Louisville, Kentucky
  - Grafton Dermatology and Cosmetic Surgery, Houma, Louisiana
  - Delricht Research, New Orleans, Louisiana
  - Washington University, St Louis, Missouri
  - Jubilee Clinical Research Inc, Las Vegas, Nevada
  - Juva Skin and Laser Center, New York, New York
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Clinical Neuroscience Solutions Cns Healthcare Memphis Research Center, Memphis, Tennessee
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Austin Institute For Clinical Research Aicr Pflugerville, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Center For Clinical Studies Webster, Webster, Texas
  - University of Utah, Murray, Utah
  - West End Dermatology Associates, Richmond, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (4):
  - Dermatology Research Institute Inc., Calgary, Alberta
  - Care Clinic, Red Deer, Alberta
  - Cca Medical Research, Ajax, Ontario
  - Lynderm Research Inc, Markham, Ontario
- Czechia (5):
  - Fakultni Nemocnice U Sv. Anny V Brne, Brno
  - Ccr Ostrava S.R.O., Ostrava
  - Ccr Czech A.S., Pardubice
  - Clintrial S.R.O., Prague
  - Krajska Zdravotni A.S. - Masarykova Nemocnice V Usti Nad Labem O.Z., Ústí nad Labem
- Germany (7):
  - Klinikum Der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Derma-Study-Center Friedrichshafen Gmbh, Friedrichshafen
  - Dermatologikum Hamburg Gemeinschaftspraxis Gbr, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Praxis Dr. Beate Schwarz, Langenau
  - Beldio Research Gmbh, Memmingen
  - Klifos - Klinische Forschung Osnabruck, Osnabrück
- Poland (2):
  - Centrum Badawcze Panaceum Agnieszka Brzezicka, Magdalena Lenkiewicz Sp. Z O.O., Elblag
  - Etg Warszawa, Warsaw
- Spain (5):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital de Manises, Manises
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: No